CLINICAL TRIAL: NCT01695915
Title: Diurnal Variation in Rectal Diameter Measured by Transabdominal Ultrasound in Healthy and Constipated Children.
Brief Title: Diurnal Variation in Rectal Diameter
Status: Completed | Type: Observational
Sponsor: Line Modin (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor-Investigator, Line Modin, Medical doctor, Vejle Hospital
Organization: Vejle Hospital (Other)
Other Study IDs: DV-Rect-UL
Record Dates: First submitted 2012-09-27; First posted 2012-09-28 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Constipation
Keywords: constipation; children; healthy; rectal diameter
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy: Transabdominal ultrasound
  Interventions: Procedure: Transabdominal ultrasound
- Constipated: Transabdominal ultrasound
  Interventions: Procedure: Transabdominal ultrasound

INTERVENTIONS:
Procedure: Transabdominal ultrasound — Transabdominal ultrasound are applied to the subjects every third hour during the study and every hour for three hours after a bowel movement.

SUMMARY:
The purpose of the study is to determine the diurnal variation of rectal diameter in healthy and constipated children using transabdominal ultrasound.

ELIGIBILITY:
Constipated Inclusion Criteria:

* Children from 4 to 12 years with previously diagnosed simple constipation defined by ROME III criteria, which at inclusion is in maintenance therapy with PEG + E and has been in treatment for at least 1 month.

Exclusion Criteria:

* Children with known organic causes of constipation, including Hirschsprungs disease, spinal and anal congenital abnormalities, previous surgery on the colon, inflammatory bowel disease, allergy and metabolic or endocrine diseases.
* Children receiving drugs known to affect bowel function during a 2 month period before initiation besides laxatives.

Healthy inclusion Criteria:

* Children between 4 and 12 years of age.

Healthy exclusion Criteria:

* Children with known organic causes of constipation, including Hirschsprungs disease, spinal and anal congenital abnormalities, previous surgery on the colon, inflammatory bowel disease, allergy and metabolic or endocrine diseases.
* Children receiving drugs known to affect bowel function during a 2 month period before initiation.
* Children with a previous history of constipation, fecal incontinence and / or urinary tract infections.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Constipated children are recruited from the outpatient clinic at Kolding pediatric department. A list of patients which have been given the diagnose constipation are drawn from the computer and reviewed. Children between 4-12 years who fulfill the Rome III criteria of constipation and have been taking PEG maintenance treatment at least 1 month, are contacted by telephone for possible participation in the study.
  Healthy participants without constipation or other diseases affecting the gastrointestinal tract were recruited among the employees of the Department of Pediatrics at Kolding Hospital.
  Written informed consent was obtained from both parents before any procedures were initiated.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Rectal diameter | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Line Modin, MD, Principal Investigator — Kolding Sygehus; Marianne Jakobsen, MD, phd, Study Director — Kolding Sygehus
Locations (1):
- Pediatric department, Kolding Hospital, Kolding, Denmark